CLINICAL TRIAL: NCT06622226
Title: A Phase 1, Open-label, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of ONO-7018 in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma (NHL) in Japan
Brief Title: A Study of ONO-7018 in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7018-03; jRCT2021240028 (Registry Identifier: Registry Identifier:)
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Tolerability (Experimental): Up to 4 dose levels will be evaluated. Eligible patients will be assigned to a dose level cohort according to a traditional 3+3 dose escalation design.
  Interventions: Drug: ONO-7018

INTERVENTIONS:
Drug: ONO-7018 — ONO-7018 tablet(s) are administered orally.

SUMMARY:
ONO-7018 is a selective inhibitor of mucosa associated lymphoid tissue protein 1 (MALT1) and is expected to exhibit antitumor activity in NHL. This study is Phase1 study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (biomarkers) and efficacy of ONO-7018 in patients with relapsed or refractory NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically/cytologically confirmed diagnosis of any of the subtypes of B-cell NHL or T-cell NHL defined below as documented by medical records and with histology based on criteria established by the World Health Organization (Swerdlow 2017)
2. Relapsed or refractory patient who is refractory or intolerant to standard therapy or for whom, in the opinion of the investigator, there is no appropriate treatment for the primary disease.
3. Patient who has measurable disease
4. Eastern Cooperative Oncology Group Performance Status 0 to 2
5. Life expectancy of at least 3 months

Exclusion Criteria:

1. Any serious or uncontrolled medical disorder that may increase the risk associated with study participation or study treatment, or interfere with the interpretation of study results
2. Patient with malignancies other than lymphoid malignancy allowed per inclusion criteria
3. Prior treatment with a MALT1 inhibitor
4. Patient is unable to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | up to 3 weeks after the first dose
  Observed toxicities will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 to assess the tolerability of ONO-7018.
Incidence, causality, and severity of Treatment emergent adverse events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Up to 28 days after the last dose
  Adverse events with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 used as a guide for the grading of severity.

SECONDARY OUTCOMES:
Plasma Concentration of ONO-7018 | up to 16 weeks after the first dose
  Plasma concentration will be assessed to evaluate Pharmacokinetics.
Maximum observed concentration (Cmax) | up to 16 weeks after the first dose
  To assess the PK profile of ONO-7018
Time to Cmax (Tmax) | up to 16 weeks after the first dose
  To assess the PK profile of ONO-7018
Area under the concentration-time curve to the end of the dosing period (AUCtau) | up to 16 weeks after the first dose
  To assess the PK profile of ONO-7018
Elimination half-life (T1/2) | up to 16 weeks after the first dose
  To assess the PK profile of ONO-7018
Predose trough concentration (Ctrough) | up to 16 weeks after the first dose
  To assess the PK profile of ONO-7018
Overall Response Rate (ORR) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by ORR will be assessed according to the response criteria for Lymphoma.
Complete response rate (CRR) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by CRR will be assessed according to the response criteria for Lymphoma.
Best overall response (BOR) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by BOR will be assessed according to the response criteria for Lymphoma.
Duration of response (DOR) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by DOR will be assessed according to the response criteria for Lymphoma.
Time to response (TTR) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by TTR will be assessed according to the response criteria for Lymphoma.
Progression-free survival (PFS) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by PFS will be assessed according to the response criteria for Lymphoma.
Overall survival (OS) | through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by OS will be assessed.
Percent change of tumor volume | through study completion, an average of 1 year
  Percent change of tumor volume will be assessed according to the response criteria for Lymphoma in order to evaluate antitumor activity of ONO-7018.
Maximum percent reduction of tumor volume | through study completion, an average of 1 year
  Maximum percent reduction of tumor volume will be assessed according to the response criteria for Lymphoma in order to evaluate antitumor activity of ONO-7018.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (6):
- Japan (6):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Shibukawa Medical Center, Shibukawa-shi, Gunma
  - Hiroshima Red Cross Hospital Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Osaka National Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No